CLINICAL TRIAL: NCT03547856
Title: A Registry Study on the "Action of Controlling Ambulatory Blood Pressure to Target in Ten Thousand Patients"
Status: Recruiting | Type: Observational
Sponsor: Yan Li (Other)
Responsible Party: Sponsor-Investigator, Yan Li, Professor of Cardiovascular Medicine, Shanghai Institute of Hypertension
Organization: Shanghai Institute of Hypertension (Other)
Other Study IDs: REACTION-ABP
Record Dates: First submitted 2018-05-02; First posted 2018-06-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Blood Pressure; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
24 hour ambulatory blood pressure (ABP) monitoring should be the first choice for diagnosis and treatment of hypertension according to European Societyof Hypertension (ESH) and the European Society of Cardiology (ESC) guideline on ambulatory blood pressure monitoring. Finally, we should promote the clinical application of 24 hour ambulatory blood pressure monitoring to greatly improve the management level of hypertension in China and effectively reduce the risk caused by hypertension in the population.

Information of hypertensive patients with ambulatory blood pressure monitoring was prospectively registered nationwide,and then to investigate whether there was difference in cardiovascular prognosis according to the control of ABP.

DETAILED DESCRIPTION:
Hypertension is the most common cardiovascular disease, and it is a fatal disease causing stroke, myocardial infarction and heart failure. Effective blood pressure management can greatly reduce the incidence of cardiovascular and cerebrovascular events. The control rate of hypertension in China is very severe. A national survey in 2002 showed that the control rate for hypertension was 6.1%. Another latest survey showed that among the 1.7 million Chinese aged 35 to 75, the detection rate of hypertension was 37 percent, among which the awareness rate and treatment rate and control rate were 36%, 23% and 6% respectively.

Traditionally, BP in the office or clinic has been assessed with the auscultatory technique, which has survived to this day in clinical practice. Although the technique is inherently accurate, it is dependent on observer attention to detail, which is lacking, and it provides only a momentary measurement of BP, usually under circumstances that can influence the level of BP being measured. To overcome these serious methodology problems, 24 hour ambulatory blood pressure techniques has been developed.

Ambulatory blood pressure monitoring is a major innovation in the development of hypertension diagnosis, and China has more than 20-year experience in clinical application of blood pressure monitoring. It measures blood pressure in a person's daily life and finds "masked hypertension", "white coat hypertension", "isolated nocturnal hypertension", "morning hypertension" and other special hypertension types. Compared with the office blood pressure, ambulatory blood pressure can better predict the incidence of target organ damage and cardiovascular events.

Ambulatory blood pressure monitoring not only can accurately assess blood pressure level, but also evaluate the effect of hypertensive therapy. Therefore, 24 hour ambulatory blood pressure monitoring should be the first choice for diagnosis and treatment of hypertension. Finally, we should promote the clinical application of 24 hour ambulatory blood pressure monitoring to greatly improve the management level of hypertension in China and effectively reduce the risk caused by hypertension in the population.

Information of hypertensive patients with ambulatory blood pressure monitoring was prospectively registered nationwide,and then to investigate whether there was difference in cardiovascular prognosis according to the control of ABP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Clinical diagnosed hypertension with the use of antihypertensive drugs
* A 24-hour ambulatory blood pressure monitoring was performed with validated equipment.
* Willing to provide information about disease history and blood biochemical test data within 6 months.
* Sign the informed consent

Exclusion Criteria:

* Without antihypertensive drug use
* Hospitalized hypertension patients
* Non-compliant patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, and community sample
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite end point of major cardiovascular and cerebrovascular events | From date of enrollment until date of first documented event or date of death from cardiovascular and cerebrovascular events, whichever came first, assessed up to 3 years
  Composite end point of major cardiovascular and cerebrovascular events

SECONDARY OUTCOMES:
The control rate of clinic blood pressure | From date of enrollment until study completion,an average of 3 years
The control rate of 24-hour ambulatory blood pressure | From date of enrollment until study completion,an average of 3 years
the proportion of white-coat uncontrolled hypertension | From date of enrollment until study completion,an average of 3 years
the proportion of masked uncontrolled hypertension | From date of enrollment until study completion,an average of 3 years
The occurrence time of cardiovascular events in different groups | From date of enrollment until date of first documented event or date of death from cardiovascular and cerebrovascular events, whichever came first, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Principal Investigator — Shanghai Institute of Hypertension
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No